CLINICAL TRIAL: NCT04786340
Title: A Randomized, Double-blind, Placebo-controlled, Parallel, 12-week, Phase 2a Study of Topical Pirenzepine (WST-057) or Placebo in Type 2 Diabetes Mellitus Patients With Painful Peripheral Neuropathy
Brief Title: A 12-Week Study of Topical Pirenzepine or Placebo in Type 2 Diabetic Patients (T2DM) With Painful Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: WinSanTor, Inc (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WST-PZP-003; 5R44DK104512 (NIH)
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Painful Diabetic Neuropathy; Diabetes Mellitus
Keywords: Diabetes Mellitus; Type 2 DM; US; WST-057
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus | interventions — Solutions

STUDY DESIGN:
Intervention Model Description: 2:1 ratio, Active (4% WST-057 topical solution): Placebo (matching placebo solution)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each subject will be randomized by an Interactive Web Response System (IWRS). When a subject is randomized, the IWRS will assign a randomization number for each subject, corresponding to a specific treatment code. The randomization number will be automatically input into the electronic Case Report Form (eCRF) by the system. The corresponding treatment code will only be accessible to the unblinded personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo: 4 mL of matching placebo topical solution. (Placebo Comparator): The placebo solution contains the same ingredients as the active solution with the exception of the active WST-057. It is dispensed with a pump to deliver 4 mL to the calves (mid-calf sock line), ankles and the tops of both feet. Both solutions (active and placebo) are applied once-a-day for 12 weeks.
  Interventions: Drug: Placebo: WST-057 4mL topical solution
- WST-057 active: 4 mL of WST-057 (4%; 146 mg of pirenzepine free base monohydrate) topical solution (Experimental): The WST-057 is the active topical solution and contains pirenzepine free base monohydrate. It is dispensed with a pump to deliver (with 4 pumps) 4 mL to the calves (mid-calf sock line), ankles and the tops of both feet. Both solutions (active and placebo) are applied once-a-day for 12 weeks.
  Interventions: Drug: Active: WST-057 4mL (146 mg pirenzepine free base monohydrate) topical solution

INTERVENTIONS:
Drug: Active: WST-057 4mL (146 mg pirenzepine free base monohydrate) topical solution — WST-057
  Arms: WST-057 active: 4 mL of WST-057 (4%; 146 mg of pirenzepine free base monohydrate) topical solution
Drug: Placebo: WST-057 4mL topical solution — Placebo
  Arms: Placebo: 4 mL of matching placebo topical solution.

SUMMARY:
This is a 12 week, 2-arm, blinded, single-site, placebo-controlled Phase II study in subjects with Type II Diabetes and painful peripheral neuropathy.

DETAILED DESCRIPTION:
This study is designed with 4 periods: screening, baseline/day 0, outpatient treatment, and safety follow-up. Site visits take place At -30 days, -7 days, Day 0, Week 3 (phone assessment), 6, 9 (phone assessment) and 12/end of study [EOS]. There is also a Week 14 phone call for a safety review with the subject. The purpose of this early phase 2 trial is to evaluate the overall safety and tolerability of both the active topical solution and the placebo also called the 'vehicle' formulated as a topical solution that penetrates the skin of the lower legs and tops of the feet. There are also secondary and exploratory objectives to determine if this active has efficacy properties during the 12-week treatment period as hypothesized. Even though pirenzepine is approved and used for another indication systemically, the sponsor believes the active in a topical solution to be effective in treating painful peripheral neuropathy commonly found in diabetic patients.

There are both objective and subjective tests being introduced in this trial due to the unique nature of the study, and lack of defined and standardized efficacy parameters.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible to participate in the study:

1. Diagnosis of T2DM (as defined by the 2016 American Diabetes Association guidelines).
2. Male and female patients in the age range of 30 to 75 years (inclusive).
3. Diagnosis of diabetic neuropathy (as defined by the Toronto Consensus Guidelines) of at least 12 months duration in the lower extremities.
4. Provide written informed consent prior to entering the study or undergoing any study procedures.
5. Females should be either not of childbearing potential as a result of surgery or menopause (1 year after onset), or of childbearing potential and must be practicing a highly effective medically acceptable method of contraception, including abstinence; hormonal contraceptives (e.g., combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device or intrauterine system; or vasectomy (partner), for at least 1 month before the screening visit and for 1 month after the end of the study. If access or use of a highly effective medically acceptable method of contraception is not achievable, then a combination of barrier methods (e.g., male condom, female condom, cervical cap, diaphragm, contraceptive sponge) is acceptable. Eligible female subjects must also have a negative serum beta-human chorionic gonadotropin at the screening visit.
6. Males must use an acceptable form of contraception (e.g., male condom with diaphragm, male condom with cervical cap, or male condom in association with spermicide).
7. Prior 24 hrs VAS for pain and/or altered sensations on lower extremities > 30 mm (0 mm = no pain-100 mm = very severe pain) at screening.
8. Participating subjects must be reliable, willing, and able to cooperate with all study procedures, including the following:

   * Return for study visits on the required dates
   * Be physically able to inspect calves, tops of ankles, and soles of feet for wounds, infections, or other anomalies, and be able to self-administer the investigational drug to calves and top surface of feet.
   * Be able to accurately and reliably report symptoms (including treatment-emergent signs and symptoms).
   * Take study drug as required by protocol.
9. Be on stable glycemic control with standard of care diabetic therapies (≥3 months prior to screening). This includes diet and exercise alone or in association with oral or injectable anti-diabetic drugs (monotherapy or combinations) that are not anticipated to change during the course of the study, except if medically required.
10. Be on stable nonpharmacological pain treatment for at least 4 weeks prior to screening and remain on this stable treatment throughout the study (unless otherwise directed by a physician). Nonpharmacologic pain treatment includes the following: relaxation/hypnosis, physical or occupational therapy, counseling, etc. Episodic or periodic treatments, such as monthly injections for treatment of pain (e.g. local anesthetics) or trans electrical nerve stimulation will not be permitted.
11. Regular and stable use of pharmacological pain treatment (less than or equal to 30 mg morphine equivalent) for at least 8 weeks prior to screening.
12. General health status must be acceptable for participation in this 12-week clinical study, with no hospitalizations for medical conditions within 12 weeks before and during screening per judgment of the Investigator. Any question regarding eligibility will be addressed with the medical monitor.
13. Fluency (oral and written) in the language in which the standardized tests will be administered.

Exclusion:

Subjects who meet any of the following exclusion criteria will be excluded from participating in the study:

1. Severe neuropathy as determined by a UENS score > 24 at screening
2. Proliferative retinopathy or maculopathy requiring acute treatment.
3. Requiring dialysis.
4. Impaired liver function, defined as aspartate aminotransferase or alanine aminotransferase > 3 times the upper limit of normal.
5. Presence of clinically significant peripheral or autonomic neuropathy that is clearly of nondiabetic origin.
6. Prior week VAS for pain and/or altered sensations on lower extremities < 30 mm (0 mm = no pain-100 mm = very severe pain) at screening.
7. Local (topical) anesthetics or analgesics including lidocaine, capsaicin, cannabinoid (CBD) oil/products or compounded topical pharmaceutical agents.
8. Uncontrolled treated/untreated hypertension (systolic blood pressure [BP] > 180 or diastolic BP > 100 at screening).
9. Amputations of lower extremities or presence of foot ulcers.
10. Clinically significant active macrovascular disease, including myocardial infarction or cerebrovascular event within the past 6 months.
11. Uncontrolled or untreated hypothyroidism.
12. Active and/or systemic infections (e.g., HIV, hepatitis, tuberculosis, syphilis), or a history of severe infection during the 30 days prior to screening.
13. Evidence of severely immunocompromised status.
14. Major surgical procedure during the 90 days prior to screening.
15. Diagnosis and/or treatment of malignancy (except for basal cell or squamous cell skin cancer, in-situ carcinoma of the cervix, or in-situ prostate cancer) within the past 5 years.
16. Clinically significant gastric emptying abnormality (e.g., severe gastroparesis).
17. Urinary retention or an enlarged prostate.
18. Uncontrolled glaucoma.
19. Other clinically significant, active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, genitourinary, endocrine, rheumatologic or hematological system that, in the opinion of the Investigator, would compromise the subject's participation in the study, might confound the results of the study, or pose additional risk in administering the study drug.
20. New treatment with (< 3 months) vitamins and supplements at the discretion of the PI.
21. Known or suspected history of alcohol or substance abuse (a stable and regular use of medical marijuana is acceptable).
22. Mental incapacity, unwillingness, or language barrier precluding adequate understanding of or cooperation with the study.
23. Women of childbearing potential who are pregnant, breast-feeding, or intend to become pregnant. Women of childbearing potential must have a negative pregnancy test at screening and must agree to use adequate contraceptive methods during the study and for 1 additional menstrual cycle following the end-of treatment visit (see inclusion criterion 5).
24. History of allergy or sensitivity to anticholinergics or any of the components of the investigational product formulations.
25. Known allergy or hypersensitivity to pirenzepine or another component of the investigational product.
26. History of sensitive skin, as defined by a requirement to use soap and skin products formulated for "sensitive skin," as determined by the Investigator.
27. Currently taking any medicines to treat overactive bladder (anticholinergic agents, such as Gelnique), or antispasmodics.
28. Failure or inability to perform screening or baseline assessments.
29. Patients with any condition that could potentially interfere with the conduct of the study or confound efficacy evaluations, including the following as specified in numbers 30 through 36 below:
30. Pain or neuropathy from another cause (including central pain, radiculopathy, painful arthritis, autoimmune and inflammatory diseases including rheumatoid arthritis, lupus, Sjogren's syndrome, vasculitic disorders such as periarteritis nodosa, Churg-Strauss, etc., celiac disease, Crohn's disease, ulcerative colitis, spondyloarthropathies, sarcoidosis, etc.) at the discretion of the PI.
31. Skin or soft-tissue lesions in the dosing area (calves, ankles and tops of feet) affected by neuropathy that are painful or could alter sensation.
32. Exposure to an experimental drug, experimental biologic, or experimental medical device within 3 months before screening.
33. Any open wound(s) and/or sunburn(s) in the dosing area. Subjects who have a wound and/or sunburn at screening that is anticipated to resolve before day -1 can be enrolled.
34. History of a serious skin disease (as determined by the Investigator), such as skin cancer, psoriasis, stasis dermatitis or eczema.
35. Receipt of a tattoo in the dosing area within 12 months of dosing.
36. Known or untreated Lyme disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events as assessed by hematology and clinical pathology blood tests | 12 weeks
  Safety will be assessed by observing changes in patients' blood tests when compared to normal lab values/ranges after once daily dosing of 1 dose level of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAEv4.0 will be reported.
Incidence of Treatment Emergent Adverse Events as assessed by vital signs (blood pressure (diastolic and systolic mmHg), heart rate (beats per minute), respiratory rate (breaths per minute). | 12 weeks
  Safety will be assessed by observing changes in patients' blood tests when compared to normal lab values/ranges after once daily dosing of 1 dose level of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAEv4.0 will be reported.
Incidence of Treatment Emergent Adverse Events as assessed by ECG (measuring p wave, QRS complex, QT interval) | 12 weeks
  Safety will be assessed by observing changes in patients' blood tests when compared to normal lab values/ranges after once daily dosing of 1 dose level of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAEv4.0 will be reported.
Incidence of Treatment Emergent Adverse Events as assessed by dermal assessment (Draize score 0.0-4.0) score of skin erythema, edema pruritus and dryness score) of the dosing area | 12 weeks
  Safety will be assessed by observing changes in patients' blood tests when compared to normal lab values/ranges after once daily dosing of 1 dose level of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAEv4.0 will be reported.

SECONDARY OUTCOMES:
Utah Early Neuropathy Score (UENS) | 12 weeks
  Utah Early Neuropathy Scale (UENS) is a simple, rapid, and reproducible test targeted to detect early sensory peripheral neuropathy. It includes motor examination, pin sensation, allodynia, hyperesthesia, large-fiber sensation, and deep tendon reflexes. The minimum score is 0. The maximum score for the UENS is 42 points. A higher score indicates more severe disease.
modified Toronto Clinical Neuropathy Score (mTCNS) | 12 weeks
  Symptomatic patient reported outcome for DPN symptoms, and neurological assessment. The minimum score is 0. The maximum score for the mTCNS is 33 points. A higher score indicates more severe disease.
Norfolk Quality of Life- Diabetic Peripheral Neuropathy (Norfolk-QOL-DN) | 12 weeks
  Patient reported outcome for quality-of-life outcomes specifically for patients with DPN. The minimum score is -4. The maximum score for the Norfolk QOL-DPN is 113 points. A higher score indicates more severe impact on a patient's quality of life.
Visual Analogue Score for Pain (VAS) | 12 weeks
  Validated patient reported outcome where patients rate their pain on a scale from 0-100mm. The minimum score is 0. The maximum score is 100. A higher score indicates more intense pain.
Neuropathy Total Symptom Score-6 (NTSS-6) | 12 weeks
  A patient reported outcome focused on frequency and type of DPN pain, etc. The minimum score is 0. The maximum score for the NTSS-6 is 21.96 points. A higher score indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hansen, Study Director — WinSanTor, Inc
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.